CLINICAL TRIAL: NCT03436004
Title: Evaluation of Colonoscopy With a Specific Device for the Detection of Adenomas: Multicenter, Prospective and Randomized Study
Brief Title: Evaluation of Colonoscopy With a Specific Device for the Detection of Adenomas
Acronym: ENDOCOLES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Alberto Herreros de Tejada Echanojáuregui (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor-Investigator, Dr. Alberto Herreros de Tejada Echanojáuregui, Principal Investigator, Puerta de Hierro University Hospital
Organization: Puerta de Hierro University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ENDOCOLES
Record Dates: First submitted 2018-01-26; First posted 2018-02-19 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Colorectal Cancer; Adenoma Colon
Keywords: Colonoscopy; Adenoma; Adenoma detection rate
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma | interventions — Colonoscopy

STUDY DESIGN:
Intervention Model Description: Randomized Multicenter prospective trial with medical device
Masking Description: Concealed assignation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Colonoscopy with specific device with CE marking (Endocuff Vision)
  Interventions: Device: Colonoscopy with specific device (Endocuff Vision)
- Active Comparator (Active Comparator): Colonoscopy with standard device of the center
  Interventions: Device: Colonoscopy

INTERVENTIONS:
Device: Colonoscopy — Patients undergoing screening colonoscopy
  Arms: Active Comparator
Device: Colonoscopy with specific device (Endocuff Vision) — Patients undergoing screening colonoscopy using the Endocuff Vision device
  Arms: Experimental

SUMMARY:
Evaluation of colonoscopy with a specific device for the detection of adenomas: Multicenter, prospective and randomized study

DETAILED DESCRIPTION:
Given the discrepancy in the results of the published studies, the main objective of the present study would be to evaluate, through a multicentric design and with a sufficiently large sample of patients, if there are relevant differences in the ADR and in the MAP between the colonoscopy performed with a device specific (Endocuff visionTM) versus standard colonoscopy.

Secondarily, the number of adenomas, the number of advanced adenomas and the number of serrated lesions in both groups.

ELIGIBILITY:
Inclusion Criteria:

All patients must be adults (≥18 years), give their consent for endoscopic exploration, for the study and meet following inclusion criteria:

1. Patients with positive immunologic fecal occult blood test (IFOBT) for population screening.
2. Patients invited to an opportunistic screening colonoscopy or included regional population screening program.
3. Patients with a family history of CRC and indication of screening colonoscopy.
4. Patients with follow-up colonoscopy indication by personal history of adenomas.

Exclusion Criteria:

1. Patients with absolute contraindications for colonoscopy (suspicion of intestinal obstruction or perforation, acute diverticulitis suspected or confirmed 6 weeks before the colonoscopy, etc).
2. Symptomatic patients with indication of diagnostic colonoscopy.
3. Patients with a personal history of CRC.
4. Patients with a personal history of chronic inflammatory bowel disease (IBD).
5. Patients with a known personal history of hereditary CRC syndrome:

   I. No polyposis (Lynch syndrome). II. Polypic.
6. Patients with suspected attenuated polyposis (> 20 adenomas) with genetic diagnosis not defined.
7. Patients with total or partial colic resection.
8. Complete colonoscopy with an adequate preparation (total Boston ≥6 with at least score ≥2 per segment) in a period of less than a year
9. Pregnant or breastfeeding mothers.
10. Patients who have expressed their wish not to participate or who do not have the ability to understand and / or sign informed consent.
11. Patients with any serious and uncontrolled medical, psychological, psychiatric, geographic or social problem that could interfere with the participation of the patient in the study or not allow an adequate follow-up and adherence with the protocol and evaluation of the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1453 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate (ADR) | 1 day
  Number of adenoma detected by colonoscopy
Mean adenoma per procedure (MAP) | 1 day
  Mean of adenoma detected by patient

SECONDARY OUTCOMES:
Total number of adenomas detected by colonoscopy | 1 day
Total number of advanced adenomas detected by colonoscopy | 1 day
Total number of serrated lesions with or without detected dysplasia by colonoscopy | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Herreros de Tejada, MD, PhD, Principal Investigator — Puerta de Hierro University Hospital; Aurora Burgos, MD, Principal Investigator — La Paz University Hospital
Locations (8):
- Spain (8):
  - Department of Gastroenterology, Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Department of Gastroenterology, Hospital Universitario La Princesa, Madrid
  - Department of Gastroenterology, Hospital General Universitario Gregorio Marañón, Madrid
  - Department of Gastroenterology, Hospital Universitario Ramón y Cajal, Madrid
  - Department of Gastroenterology, Hospital Clínico San Carlos, Madrid
  - Department of Gastroenterology, Hospital Universitario 12 de Octubre, Madrid
  - Department of Gastroenterology, Hospital Universitario La Paz, Madrid
  - Department of Gastroenterology, Hospital Universitario Fundacion Alcorcon, Madrid

IPD SHARING:
Plan to Share IPD: Undecided